CLINICAL TRIAL: NCT05070884
Title: Clinical Validation of Radiomics Artificial Intelligence: Application to Breast Cancer
Brief Title: Clinical Validation of Radiomics Artificial Intelligence: Application to Breast Cancer Treatment Planning
Acronym: RADIOVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Karolinska Institutet (Other); Medical University of Gdansk (Other); Medical School University of Zagreb (Unknown); Medical University of Vienna (Other); Hacettepe University (Other); Alexander Fleming Institute (Unknown); Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: RADIOVAL
Record Dates: First submitted 2021-09-20; First posted 2021-10-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non respondants of neo treatment: those patients with no response or partial response when administered with Chemotherapy prior to sugery
  Interventions: Other: The development of new clinical AI solutions to predict treatment response to neoadjuvant chemotherapy (NAC) in breast cancer

INTERVENTIONS:
Other: The development of new clinical AI solutions to predict treatment response to neoadjuvant chemotherapy (NAC) in breast cancer — Evaluate response to neoadjuvant treatment in advanced breast cancer

SUMMARY:
RadioVal will develop and implement interoperable solutions for clinical deployment of the radiomics tools, including information, training, and communication packages for clinicians and patients, as well as standard operating procedures for the integration of radiomics in clinical oncology. With this study, we will clinically validate these solutions, by looking at their reliability for precise breast cancer diagnosis, treatment recommendation and prognosis estimate, treatment response, evaluation of residual disease and outcome prediction.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years up to 85 years old
* Individuals referred to hospitals for diagnosis of breast cancer
* Availability of radiological images: 2D mammography or 2D synthetic digital tomosynthesis, ultrasound, or magnetic resonance
* Availability of pathological report (surgical specimen)
* Availability of (Neoadjuvant) treatment allocation (scheme, duration, benefit)
* Availability of treatment response

Exclusion Criteria:

* Patient with incomplete or low-quality data (radiological, pathological or clinical)

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients treated with chemotherapy prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients non-respondents vs respondents in neoadjuvant breast cancer treatment (Estimate tumor aggressiveness) | Baseline and after neoadjuvant treatment (4-6 months)
  Proportion of patients who have complete response evaluating the target lesion according to Miller/Payne Grading system [Ogston et al., 2003]: 1A. Evaluation of target Tumor: G5 as pathological complete response, no tumor left; G4:more than 90% loss of tumor cells; G3: between 30-90% reduction in tumor cells; G2: loss of tumor <30%; G1: no reduction. 1B: Evaluating the lymph nodes: A: negative; B: lymph nodes with metastasis and without changes by chemotherapy; C: lymph nodes with metastasis with evidence of partial response, D: lymph nodes with changes attributed to response without residual infiltration. 1C: Using images to evaluated radiological response: Size and diameter in millimeters of the target lesion using RM and TC or PET/CT for extension analysis (lymph nodes and metastasis).

CONTACTS AND LOCATIONS:
Locations (8):
- Alexander Fleming, Buenos Aires, Argentina
- Medical University of Vienna, Vienna, Austria
- University of Zagreb School of Medicine, Zagreb, Croatia
- Ain Shams University, Cairo, Egypt
- Medical University of Gdansk, Gdansk, Poland
- Hospital Universitario y Politécnico La Fe de Valencia, Valencia, Spain
- Karolinska Institute, Stockholm, Sweden
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
N/D